CLINICAL TRIAL: NCT03250260
Title: The Use of 3D Surface Imaging to Simulate Outcome After Breast Conserving Therapy
Brief Title: Simulating Outcomes From Breast Conserving Surgery Using 3D Surface Imaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CCR 4660
Record Dates: First submitted 2017-06-15; First posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer Female
Keywords: 3-dimensional imaging; Breast Conserving Treatment; Simulation

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Care (No Intervention): Patient receives standard pre-operative preparation which involves a discussion in to the likely aesthetic outcome with their surgeon or specialist nurse
- 2-dimensional Portfolio (Experimental): Patient views photographs of women matched for BMI, age, and breast volume who are 1-5 years post BCT pre-operatively.
  Interventions: Other: Viewing of a 2-dimensional photographic library
- 3-dimensional simulation (Experimental): Patient pre-operatively views a simulation of their own breast of their likely outcome after BCT.
  Interventions: Other: 3-dimensional photograph with simulation

INTERVENTIONS:
Other: 3-dimensional photograph with simulation — The viewing of a 3-dimensional simulation is classed as an intervention as it strays from the normal pre-operative preparation.
  Arms: 3-dimensional simulation
Other: Viewing of a 2-dimensional photographic library — The viewing of a 2-dimensional photograph library is classed as an intervention as it strays from the normal pre-operative preparation.
  Arms: 2-dimensional Portfolio

SUMMARY:
Most women with breast cancer are able to have an operation to remove the cancer while preserving the breast (breast conserving therapy, BCT). Whilst cancer control is the most important goal, appearance of the breast after surgery has been shown to affect the quality of a woman's life after treatment. This is even more relevant now that most women are surviving breast cancer.

Before surgery, women are prepared for how they will look afterwards by having a discussion with the Surgeon or Breast Care Nurse. Sometimes women are shown two dimensional (2D) (standard) photographs of other women who had a similar operation. Patients have stated that viewing photographs of other patients does not prepare them adequately for their own experience of surgery.

Three dimensional (3D) digital photography is currently being used to predict the appearance of the breasts after enlargement surgery using specialist software. The investigators intend to use a similar system to simulate a patient's appearance after BCT for cancer. The investigators believe that this will lead women to feel better prepared for their surgery, reduce stress, and lead to greater satisfaction with their breast after treatment.

This study invites women undergoing BCT to be assigned at random to one of three groups receiving standard care (discussion), a 2D photograph, or the 3D simulation before their operation. The investigators will find out whether women feel better prepared for surgery and are more satisfied with their outcome if they are shown a simulated image of how their own breasts are likely to look.

By taking 3D photographs of all study patients before and after surgery, a more accurate way to predict appearance after surgery will be developed for future patients.

DETAILED DESCRIPTION:
Women who are planning to have breast conserving therapy (BCT) (surgery and radiotherapy, BCT) will be identified via two pathways: 1) via the Multi-Disciplinary Team Meeting (MDM) or 2) the consulting clinician. At their surgical outpatient appointment, the patients will be given written information to take away and read at their convenience. After at least 24 hours a member of the study team will telephone the patient to answer any further questions and to see whether they would like to be considered for the trial. Women who wish to participate will have a face-to-face meeting arranged with one of the co-investigators.

At the face-to-face meeting the investigators will go through the study in detail and ask the participant to sign a consent form to allow themselves to be included in the trial. The investigators will make it clear that participants can withdraw at any point during the study. The investigators will answer any further questions, take a baseline 3-D surface image (this is done by a member of the study team in a closed room with a lockable door with the offer of a chaperone), and issue a BCT BREAST-Q.

BCT BREAST-Q is a questionnaire which has been designed for women with breast cancer who are undergoing BCT to look at their quality of life and satisfaction with different aspects of their treatment and outcome. It is split into two sections, one to be filled in before, and one after treatment.

At the face-to-face meeting, the participants will be randomly allocated into 3 groups by a computer so the study team are not involved in the decision. This makes sure the allocation is fair. All women will receive the standard care for BCT which involves a conversation with surgeon and specialist breast care nurse.

Group 1 will receive standard care only. Group 2 will be shown photographs of women who have had BCT by a member of the study team .

Group 3 will be shown a real time simulation of how their own breast is likely to look after BCT.

The preparation for group 2 and 3 will take place in a quiet closed room with the patient and co-investigator and a friend or relative if the patient wishes.

Next, the participants will be asked to complete a Visual Analogue Scale (VAS) which is a ten point scale ranging from worst-to-best (0-10) where the participant is asked to place a cross along the scale to rate their response to a specific question. The question "How confident are you that you know how your breasts are likely to look after treatment?" will be used at this point. This will conclude the face-to-face meeting. The investigators estimate the visit will take 30-40 minutes in total.

In summary thus far, after the face-to-face meeting all study participants will have given written consent, had a baseline 3D-SI, been randomised, received their appropriate preparation depending on the group allocation, have filled in a VAS for "How confident are you that you know how your breasts are likely to look after treatment?", and will have been issued with a BREAST-Q BCT questionnaire to fill out while they are waiting for randomisation or their simulation or to fill in at home and bring with them on the day of surgery.

The follow up plans will include 3D-SI, a further VAS for the question "How well do you think the information you were given about how your breasts are likely to look after surgery (discussion, 2D photographs, or 3D simulation) reflects how they actually look today?", and BCT BREAST-Q.

The 3D-SI will be taken at two weeks after their surgery (to coincide with the routine outpatient surgical appointment), before radiotherapy (to coincide with the first session of radiotherapy), 3 months after radiotherapy (to coincide with the routine radiotherapy out-patient check-up), 6 months after radiotherapy (this will need to be an additional appointment - parking charges will be refunded), at 12 months following treatment (to coincide with their normal follow-up mammogram appointment), and then annually for 5 years (to coincide with their routine mammogram appointments).

The BCT BREAST-Q will be administered at 3 and 12 months post radiotherapy (at the same time as the 3D-SI appointments above), and then annually for 5 years (at the routine mammography appointments).

The VAS for "How well do you think the information you were given before surgery about how your breasts are likely to look after surgery (discussion, 2D photographs, or 3D simulation) reflects how they actually look today?" will be administered at 3 and 12 months post treatment. The results from the VAS before treatment will be analysed to show whether there was a difference between treatment groups in participants' preparedness for surgery.

The results from the BCT BREAST-Q will show whether there was a difference between groups for how satisfied participants were with the information given to them about BCT, satisfaction with their breast, and overall quality of life during and after BCT.

The 3D-SIs taken after at 3 and 12 months post BCT will be used for comparison with the simulation model in order to improve and make it as realistic as possible. The investigators will use the 3D-SI at all time points to look at how the breasts change over time up until five years following BCT.

The post operative VAS will be used to see if the participants thought their preparation for treatment matched reality following BCT. The investigators used three groups in this study as simulation for BCT has never been done before so the investigators do not know what the best method of preparation will be. However, most hospitals do not have access to a 3D camera and it may be that much of the benefit in terms of patient preparation and confidence can be achieved by reviewing photographs which would be more generalisable within the NHS. Hence the investigators also need to compare standard care with being shown 2D photographs, and 2D with 3D.

The investigators will be working from one hospital (one of the biggest breast cancer centres in the UK) where 8 BCT operations per week are performed. When looking at how long it would take to recruit enough women for the study to make the results meaningful the investigators presumed that only half of the women approached would want to participate (less then our previous experience with similar trials which was more than three quarters). With this in mind the investigators calculated it would take 30 weeks to gather enough participants into the trial.

The trial will finish 5 years after the last participant has finished BCT.

ELIGIBILITY:
Inclusion Criteria:

Female patients Over 18 years Planned for unilateral breast conserving surgery at RMH Planned to receive adjuvant whole breast radiotherapy at RMH Willing to attend for study follow up visits.

Exclusion Criteria:

* Previous or concurrent surgery to the contralateral breast (previous breast conserving surgery, breast reduction or mastectomy)
* Previous surgery to the ipsilateral breast
* Unable to stand for long enough to have clinical photos (approximately 5 minutes)
* Unable to answer the BREAST-Q questionnaire (e.g. learning difficulties)
* Visually impaired (so that they could not view a 2D/3D images)
* Pre-operatively planning to have a symmetrisation procedure after radiotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The difference between groups in the mean pre-operative Visual Analogue Scale. | preoperatively
  The mean VAS score (range: 0 -10mm) will be compared between groups. It is intended to assess preparedness for surgery of the women in each of the three arms. Patient scores in answer to the question "How confident are you that you know how your breasts are likely to look after treatment?" will be measured for each patient following randomisation and completion of their pre-operative preparation depending on study group.

SECONDARY OUTCOMES:
The differences in post-operative 'Satisfaction with Information' scores between the 3 groups | preoperatively , 3 months and 12 months
  The difference in mean BCT BREAST-Q 'satisfaction with information' domain scores will be compared between groups at 3 and 12 months post BCT. The mean of the 4 most relevant scales within the 'satisfaction with information' domain (6i-6l) will be compared between groups separately.
The difference in 'satisfaction with breasts' score pre and post-operatively between the 3 groups. | preoperatively , 3 months and 12 months
  The mean difference between pre and post operative score for satisfaction with breasts will be compared between groups at 3 and 12 months.
The difference in 'Quality of Life' score pre and post-operatively between the 3 groups. | preoperatively , 3 months and 12 months
  The mean difference between pre and post operative score for 'quality of life' will be compared between groups at 3 and 12 months.

OTHER OUTCOMES:
The difference in post-operative VAS score between groups. | 3 months and 12 months
  The mean VAS (0-10mm) will be compared between groups at 3 and 12 months post treatment. The VAS will relate to the question: "How well do you think the information you were given before your surgery about how your breasts are likely to look after surgery (discussion, 2D photographs, or 3D simulation) reflects how they actually look today?"
The differences in linear mammometrics between 3D-Simulation and post operative reality | 3 months and 12 months
  Linear mammometrics will be compared between the simulation and the actual outcome captured on 3D-SI at 3 and 12 months in order to assess how accurate the simulation was to reality. All measurements will be represented as percentage change from the simulation to the post-operative 3D-SI (simulation/3D-SI x100).
The differences in volume measurement between 3D-Simulation and post operative reality | 3 months and 12 months
  Volume measurements will be compared between the simulation and the actual outcome captured on 3D-SI at 3 and 12 months in order to assess how accurate the simulation was to reality. All measurements will be represented as percentage change from the simulation to the post-operative 3D-SI (simulation/3D-SI x100).
The differences in surface asymmetry between 3D-Simulation and post operative reality | 3 months and 12 months
  Surface asymmetry measurements will be compared between the simulation and the actual outcome captured on 3D-SI at 3 and 12 months in order to assess how accurate the simulation was to reality. All measurements will be represented as percentage change from the simulation to the post-operative 3D-SI (simulation/3D-SI x100).
The differences in skin colour between 3D-Simulation and post operative reality | 3 months and 12 months
  Skin colour values will be compared between the simulation and the actual outcome captured on 3D-SI at 3 and 12 months in order to assess how accurate the simulation was to reality. Colours values will be presented as absolute numbers (continuous data).
The change in linear mammometrics over time. | 5 years
  Linear mammometrics will be compared using 3D-SIs of the operated and non-operated breast over time. The measurements will be represented as percentage change over time.
The change in volumes over time. | 5 years
  Volumes will be compared using 3D-SIs of the operated and non-operated breast over time. The measurements will be represented as percentage change over time.
The change in surface asymmetry over time. | 5 years
  Surface asymmetry will be compared using 3D-SIs of the operated and non-operated breast over time. The measurements will be represented as percentage change over time.
The change in colour values over time. | 5 years
  Colour values will be compared using 3D-SIs of the operated and non-operated breast over time. The measurements will be represented as percentage change over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Marsden Hospital, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Godden AR, Micha A, Wolf LM, Pitches C, Barry PA, Khan AA, Krupa KDC, Kirby AM, Rusby JE. Three-dimensional simulation of aesthetic outcome from breast-conserving surgery compared with viewing photographs or standard care: randomized clinical trial. Br J Surg. 2021 Oct 23;108(10):1181-1188. doi: 10.1093/bjs/znab217. PMID 34370833